CLINICAL TRIAL: NCT02955160
Title: A Phase 1, Randomized, Controlled, Observer-blinded Trial To Evaluate The Safety And Immunogenicity Of A Multivalent Pneumococcal Conjugate Vaccine In Healthy Adults Aged 18 To 49 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B7471001
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — Vaccines, Combined

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multivalent (Experimental): Pneumococcal conjugate vaccine
  Interventions: Biological: Multivalent
- Tdap (Active Comparator): Tetanus, diphtheria, and pertussis vaccine
  Interventions: Biological: Tdap

INTERVENTIONS:
Biological: Multivalent — Pneumococcal conjugate vaccine
  Arms: Multivalent
Biological: Tdap — Tetanus, diphtheria, and pertussis vaccine
  Arms: Tdap

SUMMARY:
This is a Phase 1 first-in-human, randomized, controlled, observer-blinded study with a 2-arm parallel design. Healthy adults aged 18 to 49 years of age with no history of pneumococcal vaccination will be randomized equally to receive either a single intramuscular dose of multivalent pneumococcal conjugate vaccine or a licensed tetanus, diphtheria, acellular pertussis combination vaccine (Tdap) (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults 18 to 49 years of age.
2. Healthy adults determined by medical history, physical examination, laboratory screening, and clinical judgment to be eligible for the study.
3. Negative serum pregnancy test for all female subjects who are of childbearing potential.

Exclusion Criteria:

1. Baseline laboratory test results outside of the normal reference range considered clinically significant.
2. History of severe adverse reaction and/or severe allergic reaction (eg, anaphylaxis) associated with a vaccine.
3. History of culture-proven invasive disease caused by S pneumoniae.
4. Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.
5. Vaccination with diphtheria-, pertussis-, or tetanus-containing vaccine(s) from 12 months before investigational product administration, or planned receipt through study participation.
6. Male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study participation and for at least 6 months after the last dose of investigational product.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects reproting prompted local reactions within 14 days after vaccination (redness, swelling. limitation of arm movement, and pain at injection site). | Day 15
Percentage of subjects reporting prompted systemic events within 14 days after vaccination (fever, headache, fatigue, chills, rash, decreased appetite, nausea/vomiting, new muscle pain, aggravated muscle pain, new joint pain, and aggravated joint pain). | Day 15
Percentage of subjects reporting adverse events (AEs) within 1 month after vaccination. | 1 month after vaccination
Percentage of subjects with clinical laboratory abnormalities after vaccination. | Day 6
Percentage of subjects reporting serious adverse events (SAEs) and newly diagnosed chronic medical conditions (NDCMCs) within 6 months after vaccination. | 6 months after vaccination

SECONDARY OUTCOMES:
Pneumococcal serotype-specific opsonophagocytic activity (OPA) geometric mean titers (GMTs) measured 1 month after vaccination. | 1 month after vaccination
Pneumococcal serotype-specific OPA geometric mean fold rises (GMFRs) measured from before vaccination to 1 month after vaccination. | 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7471001&StudyName=A%20Phase%201%2C%20Randomized%2C%20Controlled%2C%20Observer-blinded%20Trial%20to%20Evaluate%20the%20Safety%20and%20Immunogenicity%20of%20a%20Multivalent%20Pneumococcal%20Conjugate%20Vaccine%20in%20Healthy%20Adults%20Aged%2018%20to%2049%20Years
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7471001&StudyName=A+Phase+1%2C+Randomized%2C+Controlled%2C+Observer-blinded+Trial+To+Evaluate+The+Safety+And+Immunogenicity+Of+A+Multivalent+Pneumococcal+Conjugate+Vaccine+In+Healthy+Adults+Aged+18+To+49+Years